CLINICAL TRIAL: NCT06038708
Title: BIO|Sync-HUTT: Head-up Tilt Test in Patients With Reflex Syncope and Asystolic Response Who Received a Dual-chamber Pacemaker With the Closed Loop Stimulation (CLS) and Participated in the BIOSync Trial
Brief Title: Head-up Tilt Test in Patients With Reflex Syncope and Asystolic Response Who Received a Dual-chamber Pacemaker With the Closed Loop Stimulation (CLS) and Participated in the BIOSync Trial
Acronym: BIO|Sync-HUTT
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: BA117
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Syncope; Syncope, Vasovagal
Keywords: Syncope; Head-up Tilt Test; Closed Loop Stimulation; CLS
MeSH Terms: conditions — Syncope; Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore changes in patients' hemodynamic parameters during the Head-Up Tilt Test ("HUTT") and their timing with respect to onset of the Closed Loop Stimulation (CLS) pacing. This study aims to add knowledge to better understand the mechanisms underlying recurrent syncopal events and optimal pacing programming.

DETAILED DESCRIPTION:
The 2021 European Society of Cardiology guidelines recommend cardiac pacing in patients aged >40 years with tilt-induced asystolic reflex syncope (class I, level of evidence A). The recommendation relies on recent results from the multicentre, randomised, double-blinded, parallel-design BIOSync trial (NCT02324920). The BIOSync study provided evidence of benefit of dual chamber pacing in patients with tilt-induced reflex syncope and confirmed the role of Head-up Tilt Table (HUTT) test as a diagnostic method for cardiac pacing in reflex syncope. The Closed Loop Stimulation (CLS) is able to measure changes in intracardiac impedance during the systolic phase of each cardiac cycle which are strictly correlated to the increased heart rate and right ventricular contraction speed which are usually present during the pre-syncope phase of the reflex. It was hypothesized that an early onset of CLS pacing may be triggered by the compensatory increase in heart rate to counteract vasodilation and pressure drop during the pre-syncope phase of the reflex. The BIOSync study showed a 77% reduced risk of syncope in the DDD-CLS group as compared to pacing off. The design of the BIOSync study did not allow to assess the specific effect that CLS adds to dual-chamber pacing. Despite DDD-CLS pacing, 22% of patients had syncopal recurrence in 2 years. Further investigations are therefore needed in order to reduce this failure rate. Indeed, it is still unclear whether syncopal recurrences should be ascribed to dominant vasodilation or if the CLS programming/functioning needs optimization to more adequately sustain cardiac output during reflex in these specific cases.

ELIGIBILITY:
Inclusion criteria

* Ability to understand the nature of the study.
* Willingness to provide written informed consent.
* Patients undergoing HUTT for monitoring of syncope, therapy adjustment, training or other medical reasons during ordinary follow-up, irrespective of study participation
* Patients who participated in the BIOSync study*.
* Patients with a dual-chamber pacing system equipped with the CLS algorithm. * If needed, inclusion of other patients who did not participate in the BIOSync study will be considered to complete study cohort, provided that they have already a CLS pacemaker system and fulfill the same inclusion/exclusion criteria of the BIOSync study.

Exclusion criteria

* Pregnant or breast feeding women.
* Age less than 40 years.
* Patients who after the BIOSync study participation have developed the following:

  * Any indication to pacemaker different from reflex syncope with positive HUTT response; or
  * Any classified indication to implantable defibrillator, cardiac resynchronization therapy according to current guidelines; or
  * Any cardiac dysfunctions likely leading to loss of consciousness (overt heart failure, ejection fraction <40%, myocardial infarction, diagnosis of hypertrophic or dilated cardiomyopathy, clinically significant valvular disease, sinus bradycardia <50 bpm or sinoatrial block, Mobitz I second degree atrioventricular block, Mobitz II second or third degree atrioventricular block, complete bundle-branch block).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with reflex syncope and positive cardioinhibitory response to Head-Up Tilt Test (HUTT) who had already participated in the BIOSync study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale di Bolzano - Azienda Sanitaria dell'Alto Adige, Bolzano
  - Monaldi - AORN dei Colli - Università della Campania "Luigi Vanvitelli", Napoli

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request to the corresponding author with permission of BIOTRONIK SE & Co. KG.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Russo V, Tomaino M, Parente E, Comune A, Giacopelli D, Napoli P, Gargaro A, Brignole M. Temporal relationship between haemodynamic changes and activation of closed-loop stimulation during a tilt-induced vasovagal syncope. Europace. 2024 Feb 1;26(2):euae045. doi: 10.1093/europace/euae045. PMID 38340330

RESULTS

PARTICIPANT FLOW:
Groups:
- DDD-CLS Patients: Patients with reflex syncope and positive cardioinhibitory response to Head-Up Tilt Test (HUTT) with a dual-chamber pacing system equipped with the CLS algorithm.
Period: Overall Study
Arm/Group | DDD-CLS Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 20

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate [Bpm] at Specific Time-points During Head-up Tilt Test (HUTT) Examination
Description: Instantaneous measurement of heart rate value at specific time-points/stages during HUTT examination. Changes in Heart rate were investigated across four stages of the HUTT: baseline (Stage 1), pre-syncopal phase (Stage 2), maximum heart rate/pacing rate (Stage 3), and syncope or lowest Systolic Blood Pressure (Stage 4).
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
beats per minute
  Heart rate at baseline (Stage 1) | 70 (7)
  Heart rate at pre-syncopal phase (Stage 2) | 88 (12)
  Heart rate at maximum HR/pacing rate (Stage 3) | 105 (14)
  Heart rate at syncope or lowest Systolic Blood Pressure (Stage 4) | 95 (13)

2. Primary Outcome: Systolic Blood Pressure at Specific Time-points During Head-up Tilt Test (HUTT) Examination
Description: Instantaneous measurement of blood pressure at specific time-points during HUTT examination. Changes in Systolic blood pressure were investigated across four stages of the HUTT: baseline (Stage 1), pre-syncopal phase (Stage 2), maximum heart rate/pacing rate (Stage 3), and syncope or lowest Systolic Blood Pressure (Stage 4).
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
mmHg
  Systolic blood pressure at baseline (Stage 1) | 143 (20)
  Systolic blood pressure at pre-syncopal phase (Stage 2) | 108 (19)
  Systolic blood pressure at maximum heart rate/pacing rate (Stage 3) | 99 (21)
  Systolic blood pressure at syncope or lowest Systolic Blood Pressure (Stage 4) | 63 (17)

3. Primary Outcome: Stroke Volume [ml] at Specific Time-points During Head-up Tilt Test (HUTT)
Description: Instantaneous measurement of stroke volume at specific time-points during HUTT examination
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
ml
  Stroke volume at time of maximum spontaneous heart rate | 54.6 (10.4)
  Stroke volume at time of maximum CLS pacing rate | 47 (8.4)
  Stroke volume at time of recovery of basic pacing rate or spontaneous rhythm after pacing | 77.9 (34.5)

4. Primary Outcome: Peripheral Resistance [Dyn·s/cm5] at Specific Time-points During Head-up Tilt Test (HUTT)
Description: Instantaneous measurement of peripheral resistance at specific time-points during HUTT examination
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: dyn*s/cm^5
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
dyn*s/cm^5
  Peripheral Resistance at time of maximum spontaneous heart rate | 1262.5 (377)
  Peripheral Resistance at time of maximum CLS pacing rate | 1226.2 (350.4)
  Peripheral Resistance at time of recovery of basic pacing rate or spontaneous rhythm after pacing | 1183.8 (347.3)

5. Primary Outcome: Time of Maximum Spontaneous Heart Rate
Description: Recording of a specific time-point during HUTT examination. This time was collected as hours:minutes:seconds (e.g. 00:35:34).
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 22.7 [21.6 to 24.6]

6. Primary Outcome: Time of Pacing Onset
Description: as for outcome 5
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 22.9 [22.0 to 24.4]

7. Primary Outcome: Time of Recovery of Spontaneous Rhythm After Pacing
Description: as for outcome 5
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 29.2 [26.4 to 32.5]

8. Primary Outcome: Time of Syncope
Description: as for outcome 5
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 24.0 [22.9 to 25.2]

9. Primary Outcome: Time of Tilt-down
Description: as for outcome 5
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 25.3 [23.4 to 37.6]

10. Primary Outcome: Duration of the Recovery Phase [Minutes]
Description: Interval from maximum pacing rate to basic rate or spontaneous rhythm
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 5.0 [3.3 to 8.3]

11. Primary Outcome: Slope in Heart Rate [Bpm/Minute] During the Recovery Phase
Description: Calculation of the rate of change of heart rate from the time of maximum pacing rate to the time of basic rate or spontaneous rhythm recovery
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: bpm/minute
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
bpm/minute | -6.0 (3.0)

12. Primary Outcome: Slope in Systolic Blood Pressure (mmHg Per Minute) During the Recovery Phase
Description: Calculation of the rate of change of systolic blood pressure from the time of maximum pacing rate to the time of basic rate or spontaneous rhythm recovery
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Mean (Standard Deviation); unit: mmHg per minute
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
mmHg per minute | 6.2 (11.5)

13. Post Hoc Outcome: Onset of CLS Pacing
Description: Time interval from CLS pacing onset to syncope or lowest blood pressure [minutes]
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 1.7 [1.5 to 3.4]

14. Post Hoc Outcome: Duration of CLS Pacing
Description: Total duration of CLS pacing (interval from pacing onset to recovery of basic rate or spontaneous rhythm) [minutes]
Time Frame: From the start to the end of the HUTT examination, assessed up to 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | DDD-CLS Patients
Number analyzed (Participants) | 14
minutes | 5.0 [3.3 to 8.3]

ADVERSE EVENTS:
Time Frame: 2 hours
Description: This is a study without a follow-up so the adverse event data collection process is limited in time. Specifically, the time frame of 2 hours (from enrollment to the end of the Head-up tilt test within one day) for adverse event data collection is an estimate of time needed for completion of study-related procedures and during which an adverse event may occur.
Arm/Group | DDD-CLS Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT06038708/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT06038708/SAP_001.pdf